CLINICAL TRIAL: NCT06004479
Title: Effect of Pregnancy and Lactation on Carotenoid Status and Bioactivity
Brief Title: Maternal Carotenoids Across Pregnancy Study
Acronym: MCAPS
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nancy Engelmann Moran, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-46721; 3092-51000-061-002S (Other Grant/Funding Number: US Department of Agriculture, Agricultural Research Service)
Record Dates: First submitted 2023-05-12; First posted 2023-08-22 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Healthy Nutrition; Pregnancy Related
Keywords: carotenoids; skin carotenoids; cognitive function; pregnancy nutrition; macular carotenoids

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, human milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pregnant: Adult females between 18-40 years old who have a confirmed pregnancy.
  Interventions: Other: Carotenoid Intake; Other: Serum carotenoid concentration
- Non-pregnant: Adult females between 18-40 years old who do not have a confirmed pregnancy.
  Interventions: Other: Carotenoid Intake; Other: Serum carotenoid concentration

INTERVENTIONS:
Other: Carotenoid Intake — Carotenoid intake assess by 24 hour dietary recalls
Other: Serum carotenoid concentration — Serum total carotenoid concentration

SUMMARY:
Before infants are born, they depend on their mother to provide the nutrients necessary to grow and develop, such as iron, folic acid, iodine and other vitamins and minerals. Pregnant people also rely on good nutrition to support their own health. In addition to essential nutrients, vitamins, and minerals, there are other natural components found in fruits and vegetables, called phytochemicals, that may support maternal and fetal health during pregnancy.

While more is known about the role of phytochemicals in adult health, surprisingly little is known about phytochemical nutrition during pregnancy. This study focuses on a group of phytochemicals, called carotenoids, during pregnancy.

The study will determine if and why levels of carotenoids in the body change across the course of pregnancy. Understanding carotenoid nutrition during pregnancy will improve the understanding ofnutrition needs of expectant mothers and their infants. To study these questions, both health pregnant and non-pregnant female adults will report on their dietary intake and participate in body measurements, health surveys, and carotenoid measurements of eyes, skin, and blood at time points corresponding with the first, second, and third trimesters of pregnancy as well as post-partum.

DETAILED DESCRIPTION:
What a pregnant person eats is important for their own health and the health of their infant during pregnancy and after birth. Fruits and vegetables contain colorful substances called "carotenoids" which support the nutritional needs of the pregnant person and the infant, may fight inflammation, and may even benefit the person's memory and thinking ability. A person's carotenoid status can be measured with a blood sample and with optical measurements of the skin and eye. What isn't known, is if or why a pregnant person's carotenoid status changes over the course of pregnancy and the early post-partum period, and if those changes have consequences for pregnant person's and infant's health.

The goal of this study is to better understand how and why body levels of carotenoids, change during pregnancy and the post-partum period. We will study whether these changes can be explained by pregnancy, a person's diet, and changes in body composition. We will study if changes in a female's carotenoid status are associated with changes in memory or thinking ability, levels of inflammation, and her infant's carotenoid levels.

Ultimately, this information can guide nutrition advice for future pregnant people.

This study involves 5 study visits for the pregnant or non-pregnant adult female participants with an option to enroll infants for the final, post-partum, visit. For the four follow-up visits, adult participants will have body measurements, will complete surveys, and will provide a blood sample. At the final visit, lactating participants will be asked to provide a milk sample. If enrolled, infant participants will provide an optional blood sample, have body measurements, have an optical skin measurement, and their participating adult guardian will complete an infant eating survey.

ELIGIBILITY:
Inclusion Criteria:

Pregnant group

* a pregnancy confirmed by positive pregnancy test and/or ultrasound
* pre-pregnancy BMI 18.5-29.9 kg/m^2
* can speak, read, and understand English
* agrees to take the prescribed daily prenatal multivitamin as recommended by their licensed prenatal healthcare provider throughout the study.

Non-pregnant group

* current BMI that is lean 18.5-29.9 kg/m^
* can speak, read, and understand English
* agrees to continue taking any daily multivitamins or supplements throughout the study
* consumes alcohol moderately as outlined by current guidelines.

Infants

* born at term (37 weeks gestation or more)
* if infant was one of multiple births, only one sibling may be enrolled.

Exclusion Criteria:

* Metabolic, kidney, liver, digestive, or malabsorptive disorders with special dietary recommendations for the adult female or infant
* currently uses tobacco, or drugs; consumes alcohol beyond current recommendations (zero in pregnancy, 1 drink daily average for non-pregnant)
* adult female currently taking any isolated carotenoid supplements or high carotenoid (>2 mg/d) supplements
* adult female currently consumes an exclusively vegan or vegetarian diet
* adult female uses medications that interfere with dietary fat absorption
* adult female has history of endocrine disorders requiring hormone administration (with the exception of medically managed hypothyroidism).
* pregnant adult female has been informed by her doctor that she will need to take hormones during her pregnancy
* adult female has current vision condition or disease that prevents them from seeing clearly regardless of corrective lenses.
* adult female is currently lactating at enrollment.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults are recruited from the community of the greater Houston, TX metropolitan area.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Serum Total Carotenoid Concentrations - 1st Trimester Equivalent | 1st Trimester Equivalent: 8 weeks 0 days-13 weeks 6 days gestation (Week 0 if non-pregnant)
  Sum of all major carotenoid species in serum collected from fasting participant.
Serum Total Carotenoid Concentrations - 2nd Trimester Equivalent | 2nd Trimester Equivalent: 22 weeks 0 days-23 weeks 6 days gestation (or week 11-12 if non-pregnant)
  Sum of all major carotenoid species in serum collected from fasting participant.
Serum Total Carotenoid Concentrations - 3rd Trimester Equivalent | 3rd Trimester Equivalent: 32 weeks 0 days -33 weeks 6 days weeks gestation (week 22-23 if non-pregnant)
  Sum of all major carotenoid species in serum collected from fasting participant.
Serum Total Carotenoid Concentrations - Post-partum | Post-partum Equivalent: 7 weeks 0 days - 8 weeks 6 days post-partum (weeks 36-37 if non pregnant)
  Sum of all major carotenoid species in serum collected from fasting participant.

SECONDARY OUTCOMES:
Skin Carotenoid Concentrations - 1st Trimester Equivalent | 1st Trimester Equivalent: 8 weeks 0 days -13 weeks 6 days gestation (Week 0 if non-pregnant)
  Skin carotenoid score measured by pressure-mediated reflection spectroscopy
Macular pigment optical density - 1st Trimester Equivalent | 1st Trimester Equivalent: 8 weeks 0 days - 13 weeks 6 days gestation (Week 0 if non-pregnant)
  Macular pigment optical density measured by heterochromatic flicker photometry
Skin Carotenoid Concentrations - 2nd Trimester Equivalent | 2nd Trimester Equivalent: 22 weeks 0d - 23 weeks 6 days gestation (or week 11-12 if non-pregnant)
  Skin carotenoid score measured by pressure-mediated reflection spectroscopy
Macular pigment optical density - 2nd Trimester Equivalent | 2nd Trimester Equivalent: 22 weeks 0 days - 23 weeks 6 days gestation (or week 11-12 if non-pregnant)
  Macular pigment optical density measured by heterochromatic flicker photometry
Skin Carotenoid Concentrations - 3rd Trimester Equivalent | 3rd Trimester Equivalent: 32 weeks 0 days - 33 weeks 6 days weeks gestation (week 22-23 if non-pregnant)
  Skin carotenoid score measured by pressure-mediated reflection spectroscopy
Macular pigment optical density - 3rd Trimester Equivalent | 3rd Trimester Equivalent: 32 weeks 0 days -33 weeks 6 days weeks gestation (week 22-23 if non-pregnant)
  Macular pigment optical density measured by heterochromatic flicker photometry
Skin Carotenoid Concentrations - Post-partum Equivalent | Post-partum Equivalent: 7 weeks 0 days - 8 weeks 6 days post-partum (weeks 36-37 if non pregnant)
  Skin carotenoid score measured by pressure-mediated reflection spectroscopy
Macular pigment optical density - Post-partum Equivalent | Post-partum Equivalent: 7 weeks 0 days - 8 weeks 6 days post-partum (weeks 36-37 if non pregnant)
  Macular pigment optical density measured by heterochromatic flicker photometry

OTHER OUTCOMES:
Subjective memory function (MAC-Q Score) - 1st Trimester Equivalent | 1st Trimester Equivalent: 8 weeks 0 days-13 weeks 6 days gestation(Week 0 if non-pregnant)
  Subjective memory function assessed by MAC-Q
Subjective memory function (MAC-Q Score) - 2nd Trimester Equivalent | 2nd Trimester Equivalent: 22 weeks 0 days - 23 weeks 6 days gestation (or week 11-12 if non-pregnant)
  Subjective memory function assessed by MAC-Q
Subjective memory function (MAC-Q Score) - 3rd Trimester Equivalent | 3rd Trimester Equivalent: 32 weeks 0 days - 33 weeks 6 days weeks gestation (week 22-23 if non-pregnant)
  Subjective memory function assessed by MAC-Q
Subjective memory function (MAC-Q Score) - Post-partum Equivalent | Post-partum Equivalent: 7 weeks 0 days - 8 weeks 6 days post-partum (weeks 36-37 if non pregnant)
  Subjective memory function assessed by MAC-Q
Serum IL-6 - 1st Trimester Equivalent | 1st Trimester Equivalent: 8 weeks 0 days - 13 weeks 6 days gestation (Week 0 if non-pregnant)
  Serum concentrations of IL-6
Serum IL-6 - 2nd Trimester Equivalent | 2nd Trimester Equivalent: 22 weeks 0 days-23 weeks 6 days gestation (or week 11-12 if non-pregnant)
  Serum concentrations of IL-6
Serum IL-6 - 3rd Trimester Equivalent | 3rd Trimester Equivalent: 32 weeks 0 days-33 weeks 6 days gestation (week 22-23 if non-pregnant)
  Serum concentrations of IL-6
Serum IL-6 - Postpartum Equivalent | Post-partum Equivalent: 7 weeks 0 days - 8 weeks 6 days post-partum (weeks 36-37 if non pregnant)
  Serum concentrations of IL-6
Serum hsCRP - 1st Trimester Equivalent | 1st Trimester Equivalent: 8 weeks 0 days-13 weeks 6 days gestation (Week 0 if non-pregnant)
  Serum concentrations of high sensitivity C-reactive protein
Serum hsCRP - 2nd Trimester Equivalent | 2nd Trimester Equivalent: 22w0d-23w6d gestation (or week 11-12 if non-pregnant)
  Serum concentrations of high sensitivity C-reactive protein
Serum hsCRP - 3rd Trimester Equivalent | 3rd Trimester Equivalent: 32 weeks 0 days-33 weeks 6 days gestation (week 22-23 if non-pregnant)
  Serum concentrations of high sensitivity C-reactive protein
Serum hsCRP - Postpartum Equivalent | Post-partum Equivalent: 7 weeks 0 days-8 weeks 6 days post-partum (weeks 36-37 if non pregnant)
  Serum concentrations of high sensitivity C-reactive protein
Serum sTNFr-II - 1st Trimester Equivalent | 1st Trimester Equivalent: 8 weeks 0 days-13 weeks 6 days gestation (Week 0 if non-pregnant)
  Serum concentrations of sTNFr-II
Serum sTNFr-II - 2nd Trimester Equivalent | 2nd Trimester Equivalent: 22 weeks 0 days-23 weeks 6 days gestation (or week 11-12 if non-pregnant)
  Serum concentrations of sTNFr-II
Serum sTNFr-II - 3rd Trimester Equivalent | 3rd Trimester Equivalent: 32 weeks 0 days-33 weeks 6 days gestation (week 22-23 if non-pregnant)
  Serum concentrations of sTNFr-II
Serum sTNFr-II - Post-partum Equivalent | Post-partum Equivalent: 7 weeks 0 days - 8 weeks 6 days post-partum (weeks 36-37 if non pregnant)
  Serum concentrations of sTNFr-II
Serum TNF-alpha- 1st Trimester Equivalent | 1st Trimester Equivalent: 8 weeks 0 days -13 weeks 6 days gestation (Week 0 if non-pregnant)
  Serum concentrations of sTNF-alpha
Serum TNF-alpha- 2nd Trimester Equivalent | 2nd Trimester Equivalent: 22 weeks 0 days-23 weeks 6 days gestation (or week 11-12 if non-pregnant)
  Serum concentrations of sTNF-alpha
Serum TNF-alpha- 3rd Trimester Equivalent | 3rd Trimester Equivalent: 32 weeks 0 days - 33 weeks 6 days gestation (week 22-23 if non-pregnant)
  Serum concentrations of sTNF-alpha
Serum TNF-alpha- Post-partum Equivalent | Post-partum Equivalent: 7 weeks 0 days - 8 weeks 6 days post-partum (weeks 36-37 if non pregnant)
  Serum concentrations of sTNF-alpha
Infant serum carotenoid concentration | 7 weeks 0 days - 8 weeks 6 days post-partum
  Serum total carotenoid concentration in 7-8 week old infants
Infant serum carotenoid concentration | Post-partum: 7 weeks 0 days - 8 weeks 6 days post-partum
  Serum total carotenoid concentration in 7-8 week old infants

CONTACTS AND LOCATIONS:
Locations (1):
- USDA/ARS Children's Nutrition Research Center, Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided